CLINICAL TRIAL: NCT02287454
Title: Integrative Group-based Cognitive Rehabilitation Efficacy in Multiple Sclerosis: a Randomized Clinical Trial
Brief Title: Integrative Group-based Cognitive Rehabilitation Efficacy in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSMC-002-UD
Record Dates: First submitted 2014-10-22; First posted 2014-11-10 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis, cognitive rehabilitation, REHACOP
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive remediation program: REHACOP (Experimental): Cognitive rehabilitation program (REHACOP) including intervention in: attention, memory, processing speed, language, executive functioning and social cognition during 3 months, 3 times per week
  Interventions: Other: cognitive remediation program: REHACOP
- Control group (No Intervention): No intervention was administered.

INTERVENTIONS:
Other: cognitive remediation program: REHACOP — Specifically, REHACOP group remediation with MS patients consisted of: four weeks training attention (sustained, selective, alternating and divided attention); three weeks focused on learning and memory (the stimulation of verbal and visual memory was combined with learning and compensatory strategies, working memory was also trained); three weeks exercising executive functioning (development, planning and attainment of objectives); three weeks focused on language (verbal fluency, syntax, grammar, vocabulary and comprehension); and one week training social cognition (social reasoning, theory of mind and moral dilemmas).
  Arms: Cognitive remediation program: REHACOP

SUMMARY:
The study design was a parallel-group randomized trial with equal randomization. Recruitment and enrollment were conducted between January 2013 and March 2013. At base-line, cognitive data was collected. Afterwards, the participants were randomly allocated to either the REHACOP group or the Control group. During 3 months the intervention with REHACOP program took place and at follow-up patients were again re-evaluated to evaluate the change in cognitive measure. Post-treatment assessment (finished by July 2013) was performed within the first week after completing the intervention. Optional enrollment in pre-post neuroimaging will also allow us to look at changes in the brain.

Objective: To examine the efficacy of an integrative cognitive training program (REHACOP) to improve cognition of patients with Multiple Sclerosis (MS).

DETAILED DESCRIPTION:
Assessment protocol:

Patients underwent an extensive neuropsychological battery including test of attention, working memory, processing speed, verbal memory (learning and recall), verbal fluency and executive functioning. Sustained attention was measured using the Brief Test of Attention. For working memory, the Backward Digits subtest of the Weschler Adult Intelligence Scale III was used. Processing speed was assessed through the Symbol Digit Modalities Test, the three and six letter version of the Salthouse Perceptual Comparison Test and the Trail Making Test A. Verbal memory was determined based on the Hopkins Verbal Learning Test , learning and long-term recall performance. For verbal fluency, the Category (animals and supermarket) and Letter (P) Word Fluency Test from the Calibrated Ideational Fluency Assessment were utilized . Executive functioning was calculated by the word-color and interference scores of the Stroop Word-Color Test.

Additionally, several test and scales were administered. The Expanded Disability Status Scale was used for rating the degree of neurologic impairment. Premorbid IQ was tested by The Accentuation Reading Test. Cognitive reserve was estimated with the Cognitive Reserve Questionnaire. The 15-item Geriatric Depression Scale was included to assess patients´ depressive symptoms. The Fatigue Severity Scale and the mental fatigue Visual Analogue Scale were included to evaluate physical and mental fatigue, respectively.

Description of the intervention:

REHACOP is a structured program using paper-pencil tasks and it is based on the principles of restoration, compensation and optimization with a gradually increasing level of cognitive effort and demand. REHACOP trains different cognitive domains, such as attention, memory, processing speed, language, executive functioning and social cognition. Additionally, the program includes one unit related to functional outcome: activities of daily living. REHACOP includes up to 300 different tasks hierarchically organized into at least three levels of difficulty and subtypes of abilities. Several tasks are timed, so processing speed is trained throughout various modules. Once a basic cognitive strategy has been trained and well acquired, the therapist transitions the program to the next level. The program format allows for either individual or group sessions (between 5 and 8 patients per group), although for the purpose of this study, group sessions were chosen. In this study, two psychologists conducted the REHACOP group attending 60-minute-long sessions 3 days per week at Multiple Sclerosis Association of Biscay (ADEMBI) (four groups). Specifically, REHACOP group remediation with MS patients consisted of: Attention unit (4 weeks) training sustained, selective, alternant and divided attention; Memory unit (3 weeks) focusing on visual and verbal learning, recall and recognizing memory, as well as in working memory; Language unit (3 weeks) including verbal fluency, grammar, syntax, vocabulary, verbal comprehension, abstract language; Executive functions unit (2 weeks) training development, planning and attainment of objectives; and Social cognition unit (1 week) exercising theory of mind, social reasoning and moral dilemmas.

ELIGIBILITY:
Inclusion Criteria:

i) age 20-60 years

ii) either male or female

iii) patients with relapsing-remitting, secondary progressive or primary progressive MS

Exclusion criteria:

i) presence of dementia

ii) have suffered an exacerbation during the previous month to the cognitive assessment

iii) being treated with corticosteroids

iv) presence of other neurological disorder

v) history of stroke or traumatic brain injury resulting in more than 30 minutes loss of consciousness

vi) presence of psychiatric disorders

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in attention after receiving cognitive rehabilitation treatment | 3 months
  Attention was measured using the Brief Test of Attention (BTA).
Change in working memory after receiving cognitive remediation treatment | 3 months
  Working memory was measured using the Backward Digits (BD) subtest of the Wechsler Adult Intelligence Scale III.
Change in processing speed after receiving cognitive remediation treatment | 3 months
  Processing speed was measured using a composite score which included the Symbol Digit Modalities Test (SDMT), the three and six letter version of the Salthouse Perceptual Comparison Test (PCT) and the Trail Making Test A (TMTA).
Change in verbal memory after receiving cognitive remediation treatment | 3 months
  Verbal memory was measured using The Hopkins Verbal Learning Test - Revised (HVLT-R).
Change in verbal fluency after receiving cognitive remediation treatment | 3 months
  Verbal fluency was measured using the Calibrated Ideational Fluency Assessment (CIFA).
Change in executive functioning after receiving cognitive remediation treatment. | 3 months
  Executive functioning was measured with the Stroop Color-Word Test.

CONTACTS AND LOCATIONS:
Overall Officials: Naroa Ibarretxe-Bilbao, Doctor, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, Bilbao, Biskai, Spain